CLINICAL TRIAL: NCT01849315
Title: Effects of an Empirically-Based Physical Activity Intervention on Chronic Disease Risk Factors in Children
Brief Title: Effects of Physical Activity on Disease Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, Cheryl Howe, Assistant Professor, Ohio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12F011
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Sedentary intervention
  Interventions: Behavioral: AKIDS II
- AKIDS II (Active Comparator): Physically active group
  Interventions: Behavioral: AKIDS II

INTERVENTIONS:
Behavioral: AKIDS II — Physically active intervention

SUMMARY:
Obesity is associated with increased risk of heart disease and diabetes (Kim et al., 2010). Appalachian children in Athens County, Ohio, experience higher rates of obesity compared to the national average (20.9% vs. 15.4%), which increases their risk of obesity-related diseases (Montgomery-Reagan, Bianco, Heh, Rettos, & Huston, 2009). Although physical activity (PA) is known to improve fitness and adiposity (Gutin & Owens, 2011; Yin et al., 2009), very little is known about the effects of PA on the progression of chronic disease risk factors (biomarkers) for obesity-related diseases in children, such as inflammatory markers, lipids, and glucose/insulin. This lack of knowledge is due to a limited understanding of the number of calories burned during children's free-play PA. This study will assess the impact of a PA program (ACT) of known energy cost on obesity-related disease markers in 2nd-4th grade children compared to a sedentary control group (SED). The study will recruit children from an after-school program in Athens County elementary schools. Baseline and posttest data will include measures of height, weight, body composition, blood pressure, and physical activity levels. Following baseline measures, children will be randomized into either the ACT or SED group for 8 weeks. The ACT group will play recess-type games previously determined to expend ≥100 calories in 30 minutes. The SED group children will play sedentary-type activities during the same time period. It is hypothesized that the ACT group children will demonstrate significant improvements in PA after 8 weeks compared to the SED group children and that these improvements will be related to positive changes in body weight and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Attends participating after school program

Exclusion Criteria:

* cardiorespiratory, metabolic, and neurological disorders and physical impairments that would prevent them from being physically active, and were not taking any medications that would affect metabolism

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Daily Physical Activity Levels | 8 weeks
  increase relative to participation in intervention

SECONDARY OUTCOMES:
body composition | 8 weeks
  attenuation in excess gains in weight and body mass index
biomarkers for cardiometabolic disease | 8 weeks
  decrease relative to intervention participation